CLINICAL TRIAL: NCT06292156
Title: tACS Treatment for Cognitive Impairments in Methamphetamine Addicts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing HuiLongGuan Hospital (Other)
Responsible Party: Principal Investigator, Xiang Yang Zhang, Professor, Beijing HuiLongGuan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CASPsy7
Record Dates: First submitted 2023-12-03; First posted 2024-03-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Methamphetamine Abuse
Keywords: Methamphetamine patients; Cognitive impairments; tACS
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Theta treatment group (Experimental): In active tACS, the target 'active' electrode was placed over the MFC and the second 'return' electrode was placed over the medial parietal cortex. 6 Hz stimulation was used and a alternating current of 2mA was applied for 30min each day(Monday-Friday) for 3 consecutive weeks.
  Interventions: Device: Theta treatment group
- Sham control group (Sham Comparator): In sham group, Sham stimulation lasted 30 s (15 s of ramp- up and 15 of ramp-down) .
  Interventions: Device: Sham control group

INTERVENTIONS:
Device: Theta treatment group — The target 'active' electrode was placed over the MFC and the second 'return' electrode was placed over the medial parietal cortex. 6 Hz stimulation was used and a alternating current of 2mA was applied for 30min each day(Monday-Friday) for 3consecutive weeks
  Arms: Theta treatment group
Device: Sham control group — Sham stimulation lasted 30 s (15 s of ramp- up and 15 s of ramp-down).
  Arms: Sham control group

SUMMARY:
1. To evaluate the cognitive function of methamphetamine Patients.
2. Investigate the pathological mechanism of methamphetamine patients from the aspects of EEG and biology;
3. The investigators investigated the effects of transcranial alternating current stimulation (tACS) on cognitive impairments in methamphetamine patients

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis diagnosis of methamphetamine use disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* None of participants had mixed use of other drugs
* None of participants had physical disability
* None of participants had acute physical or mental illness, hallucinations, acute withdrawal symptoms
* None of participants were receiving any medical treatment

Exclusion Criteria:

* Intracranial hypertension
* Cranial defects
* Tumors
* Serious physical illnesses (e.g., cardiovascular, liver, kidney, gastrointestinal disorders)
* Infectious diseases
* Immune system disorders

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) | Baseline, week 3
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS), which contains 12 subtests for calculating the index scores of delayed memory (including list recall, story recall, figure recall, and list recognition tests), attention (including digit span and coding tests), language (including picture naming and semantic fluency tests), visuospatial/constructional index (including figure copy and line orientation tasks), immediate memory (including list learning and story memory tasks), and global neuropsychological function.
ERP components associated with cognitive function | Baseline, week 3
  Investigate the ERP components associated with cognitive function of methamphetamine patients using event-related potential analysis
Condition stop signal task | Baseline, week 3
  Condition stop signal task was used to assess cognitive control function, including proactive control and reactive control.
Neural oscillations associated with cognitive function | Baseline, week 3
  Investigate the neural oscillations associated with cognitive function of methamphetamine patients using time-frequency analysis.
Functional connection of brain region associated with cognitive function | Baseline, week 3
  Investigate the functional connection of brain region associated with cognitive function of methamphetamine patients using functional connection analysis
Microstate associated with cognitive function | Baseline, week 3
  Investigate the microstate associated with cognitive function of methamphetamine patients using microstate analysis
Neural Dynamic Coding of brain region associated with cognitive function | baseline, week 3
  Investigate the functional connection of brain region associated with cognitive function of methamphetamine patients using multivariate pattern analysis
The effect of oxidative stress system on cognitive function | Baseline, week 3
  The investigators examined markers of oxidative stress related to cognitive function using bioassay.
The effect of immune system on cognitive function | Baseline, week 3
  The investigators immune indicators related to cognitive function using bioassay.
The effect of brain derived neurotrophic factor(BDNF) on cognitive function | Baseline, week 3
  The investigators BDNF indicators related to cognitive function using bioassay.
Genetic mechanism of cognitive function | Baseline, week 3
  The investigators performed comprehensive genetic testing to explore the genetic mechanism of cognitive function.

SECONDARY OUTCOMES:
Reverse learning task | Baseline, week 3
  Reverse learning task was used to access the compulsive drug using behavior of methamphetamine patients.
Beck Depression Scale | Baseline, week 3
  Beck Depression Scale was used to access degree of depression.The total score varies between 0 and 30 points, with higher scores indicating higher levels of depression.
Barrett impulse Scale | Baseline, week 3
  The scale includes three dimensions: motor impulsivity, cognitive impulsivity and unplanned impulsivity. The total score varies between 30 and 150 points, with higher scores indicating higher levels of impulsivity. High scores on the three subscales indicated hyperactivity, inattention, and lack of planning, respectively.
Degree of insomnia | Baseline, week 3
  Insomnia Severity Index was used acess the patient's insomnia.The total score varies between 0 and 28 points, with higher scores indicating higher levels of insomnia.
The Sensitivity to Punishment and Reward Questionnaire | Baseline, week 3
  The Sensitivity to Punishment and Reward Questionnaire including penalty sensitivity factor and reward sensitivity factor. The total score varies between 0 and 31 points, with higher scores indicating higher sensitivity to penalty and reward.
Visual analog scale | Baseline, week 3
  Visual analog scale（VAS） was used to acess the craving of drug on a scale of 1 to 10.A higher score indicates a higher desire for the drug
The Desires for Drug Questionnaire | Baseline, week 3
  The Desires for Drug Questionnaire (DDQ) was used to access the craving of drug, which measures three factors, including desire and intention, negative reinforcement, and control. Higher scores of drug desire and negative reinforcement indicated higher drug craving, and higher scores of control indicated better drug craving control ability.The total score on the table is equal to the sum of the scores in the three dimensions, ranging from 3 to 21 points.
Obsessive compulsive drug use scale | Baseline, week 3
  The Obsessive Compulsive Drug Use Scale (OCDUS) also measures three factors: thoughts about methamphetamine and interference, desire and control, and resistance to thoughts and intention.The higher the total score, the higher the craving. The total score varies between 13 and 65 points, with higher scores indicating higher craving.
Obsessive-compulsive inventory | Baseline, week 3
  Obsessive-compulsive inventory was evaluated the subjects' obsessive-compulsive symptoms from 6 different dimensions, including washing, forcing thoughts, storing, sorting, checking, mixing.The total score varies between 0 and 72 points, with higher scores indicating more severe obsessive-compulsive symptoms.
Thought Control Ability Questionnaire | Baseline, week 3
  Thought Control Ability Questionnaire was used to measure the ability of an individual to control unwanted and intrusive thoughts. The total score varies between 25 and 125 points, with higher indicating scores the stronger the thought control ability.
Thought Suppression Questionnaire | Baseline, week 3
  Thought Suppression Questionnaire were used to access the thought control ability. The total score varies between 15 and 75 points, with higher indicating scores the stronger the thought suppression ability.
Rumination Questionnaire | Baseline, week 3
  Rumination Questionnaire was used to access ruminate behavior.A higher total score indicates a higher tendency to ruminate. The total score varies between 22 and 88 points, with higher scores indicating higher tendency to ruminate.
Anger Rumination Questionnaire | Baseline, week 3
  Anger Rumination Questionnaire was used to access anger ruminate behavior. The total score varies between 19 and 76 points, with higher scores indicating higher tendency to anger ruminate.
Beck Anxiety Scale | Baseline, week 3
  Beck Anxiety Scale was used to access degree of anxiety.The total score varies between 0 and 63 points, with higher scores indicating higher levels of anxiety.
Emotional Regulation Difficulty Scale | Baseline, week 3
  Emotional Regulation Difficulty Scale was used to access the emotional regulation ability of methamphetamine patients.The total score varies between 36 and 180 points, with higher scores indicating the more serious the difficulty in emotion regulation and the lower the level of emotion regulation ability.
Aggressive questionnair | Baseline, week 3
  Aggressive questionnaire was used to access aggressive behavior of methamphetamine patients. The total score varies between 30 and 150 points, with higher scores indicating the more aggressive behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Xin Hua Drug Rehabilitation Center, Mianyang, China

IPD SHARING:
Plan to Share IPD: No
Data will be avaliable on request